CLINICAL TRIAL: NCT05189444
Title: The Evaluation of Triple Therapy With Vonoprazan, Amoxicillin and Bismuth for Eradication of Helicobacter Pylori: a Prospective, Multi-Center, Randomized Controlled Trial
Brief Title: The Evaluation of Triple Therapy With Vonoprazan, Amoxicillin and Bismuth for Eradication of Helicobacter Pylori
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Bin Cheng, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vonoprazan-Hp-2021
Record Dates: First submitted 2021-12-29; First posted 2022-01-12 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Helicobacter Pylori Infection
Keywords: Vonoprazan; Standard Quadruple Therapy
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; Esomeprazole; Clarithromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vonoprazan group (Experimental): Vonoprazan + Amoxicillin + Bismuth potassium citrate Drug: Vonoprazan 20mg bid Other Names: no Drug: Amoxicillin 0.75g tid Other Names: no Drug: Bismuth potassium citrate 0.22g bid Other Names: no
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin; Drug: Bismuth potassium citrate
- control group: quadruple therapy (Active Comparator): Drug: Esomeprazole 20mg bid Other Names: no Drug: Amoxicillin 1.0g bid Other Names: no Drug: Clarithromycin 0.5g bid Other Names:no Drug: Bismuth potassium citrate 0.22g bid Other Names:no
  Interventions: Drug: Esomeprazole; Drug: Amoxicillin; Drug: Clarithromycin; Drug: Bismuth potassium citrate

INTERVENTIONS:
Drug: Vonoprazan — 20mg bid
  Arms: Vonoprazan group
Drug: Amoxicillin — 0.75g tid
  Arms: Vonoprazan group
Drug: Esomeprazole — 20mg bid
  Arms: control group: quadruple therapy
Drug: Amoxicillin — 1.0g bid
  Arms: control group: quadruple therapy
Drug: Clarithromycin — 0.5g bid
  Arms: control group: quadruple therapy
Drug: Bismuth potassium citrate — 0.22g bid

SUMMARY:
The eradication rate of standard quadruple therapy has become less successful due to low compliance and high resistance to antibiotics. Therefore, it is necessary to develop new treatment strategies that increase the eradication rate and reduce adverse effects. The aim of this prospective study is to investigate the efficacy of Triple Therapy with Vonoprazan, Amoxicillin, and Bismuth for eradication of Hp, compared with standard quadruple therapy.

DETAILED DESCRIPTION:
In China, the first-line therapy to treat Helicobacter pylori (Hp) consists of a bismuth-based proton pump inhibitor (PPI) and two antibiotics for 14 days.But, eradication has become less successful due to low compliance and high resistance to antibiotics. Therefore, it is necessary to develop new treatment strategies that increase the eradication rate and reduce adverse effects. Vonoprazan is a novel potassium-competitive acid blocker more effective in suppressing acid production than proton pump inhibitors (PPIs). Several studies previously suggested that vonoprazan containing antibiotic therapy was superior to other PPI-containing therapies for Hp. Most strains of Helicobacter pylori are sensitive to amoxicillin. Bismuth salts, a topical agent, which are available in our country, have a synergistic effect on antibiotics and decrease the bacterial load. Therefore, the investigators performed a prospective, multi-center, randomized trial, to investigate the efficacy of Triple Therapy with Vonoprazan, Amoxicillin, and Bismuth for eradication of Hp, compared with standard quadruple therapy.

ELIGIBILITY:
Inclusion Criteria:

* Helicobacter pylori infected patients comfirmed by 13C/14C UBT
* age 18~65

Exclusion Criteria:

* prior Hp eradication therapy including amoxicillin and clarithromycin
* previous gastric resection
* allergic to the drugs used in this study
* previous use of proton pump inhibitors, bismuth, H2 receptor antagonist or antibiotics, probiotics within 4 weeks of the study
* Patients who were pregnant or lactating
* Patients taking NSAIDs, alcoholic or with other serious disease (e.g. hepatopathy, heart disease, nephropathy#diabete mellitus, hypertension…) effect the evaluation of this study
* Can't express the complaint correctly

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 672 (Estimated)
Dates: Start 2022-03-25 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication | 6 weeks after treatment initiation
  to investigate the efficacy of Triple Therapy with Vonoprazan, Amoxicillin and Bismuth for eradication of Hp, compared with standard quadruple therapy.

SECONDARY OUTCOMES:
Incidence of adverse events | 2 weeks and 6 weeks after treatment initiation
  to investigate the incidence of adverse events of Triple Therapy with Vonoprazan, Amoxicillin and Bismuth, compared with standard quadruple therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cheng, Doctor, Principal Investigator — Tongji Hospital; si xiong, Doctor, Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, HUST, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gunaratne AW, Hamblin H, Clancy A, Magat AJMC, Dawson MVM, Tu J, Borody TJ. Combinations of antibiotics and vonoprazan for the treatment of Helicobacter pylori infections-Exploratory study. Helicobacter. 2021 Oct;26(5):e12830. doi: 10.1111/hel.12830. Epub 2021 Jul 10. PMID 34247436
- [Result] Rokkas T, Gisbert JP, Malfertheiner P, Niv Y, Gasbarrini A, Leja M, Megraud F, O'Morain C, Graham DY. Comparative Effectiveness of Multiple Different First-Line Treatment Regimens for Helicobacter pylori Infection: A Network Meta-analysis. Gastroenterology. 2021 Aug;161(2):495-507.e4. doi: 10.1053/j.gastro.2021.04.012. Epub 2021 Apr 8. PMID 33839101
- [Result] Kiyotoki S, Nishikawa J, Sakaida I. Efficacy of Vonoprazan for Helicobacter pylori Eradication. Intern Med. 2020 Jan 15;59(2):153-161. doi: 10.2169/internalmedicine.2521-18. Epub 2019 Jun 27. PMID 31243237
- [Result] Ang TL, Ang D. Helicobacter pylori Treatment Strategies in Singapore. Gut Liver. 2021 Jan 15;15(1):13-18. doi: 10.5009/gnl19308. PMID 31875670
- [Result] Kao CY, Sheu BS, Wu JJ. Helicobacter pylori infection: An overview of bacterial virulence factors and pathogenesis. Biomed J. 2016 Feb;39(1):14-23. doi: 10.1016/j.bj.2015.06.002. Epub 2016 Apr 1. PMID 27105595